CLINICAL TRIAL: NCT02636010
Title: Phase II, Multicenter, Open Label, Clinical Trial of the Anti-PD1 Monoclonal Antibody Pembrolizumab (MK-3475) as Consolidation Therapy in Multiple Myeloma Patients With Residual Disease After Treatment
Brief Title: Pembrolizumab (MK-3475) in MM Patients With Residual Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Adknoma Health Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-PEMBRESID
Record Dates: First submitted 2015-11-25; First posted 2015-12-21 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK-3475 Pembrolizumab (Experimental): MK-3475 at a dose of 200 mg every three weeks for 1 year with a potential expansion of 1 additional year of treatment in case of clinical benefit and patient agreement
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: MK-3475

SUMMARY:
This is a national, multicenter, open label single-arm, non-comparative study that will determine the efficacy, safety and the changes in selected pharmacodynamics markers of MK-3475 monotherapy administered as consolidation therapy in MM patients who have achieved a response with a previous treatment but who still display some residual disease.

For this purpose, 20 MM patients, who have received any treatment of limited duration either at diagnosis or at first relapse, and that have achieved a good response (≥VGPR) but with persistent residual disease (that is patients in VGPR, non-stringent CR, or MRD+ sCR), will be treated with MK-3475 monotherapy administered iv at a dose of 200 mg every three weeks for 1 year, with a potential expansion of 1 additional year of treatment in case of clinical benefit and patient agreement. Efficacy, safety and pharmacodynamic parameters will be evaluated to understand the role of this monoclonal antibody in this setting.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a B cell malignancy characterized by the presence of bone marrow infiltration by clonal plasma cells that generally secrete a monoclonal component in the serum or urine. It is the second most frequent hematological malignancy, after non-Hodgkin lymphomas, and accounts approximately for a 10% of all hematological tumors and 1% of all cancers. Treatment of MM has remained substantially unchanged for some time (reviewed in with alkylating agents such as melphalan in combination with steroids being the gold standard for more than 25 years. Later on, in the 1970 decade, other drugs such as carmustine or vincristine where combined with melphalan, cyclophosphamide or steroids giving rise to the chemotherapeutic regimens; and ten years later high doses of melphalan with autologous stem cell transplantation (ASCT) where introduced into the clinical practice. All these treatment schemes resulted in an overall survival of around 30 months until 1994 with a slight improvement in the subsequent five years, probably due to the introduction of ASCT and better measures of supportive care. Finally, in the first decade of this century, some new drugs with novel mechanisms of action and clear antimyeloma activity have been discovered and approved. In this regard, several studies have demonstrated the activity of the proteasome inhibitor bortezomib and the immunomodulatory agents thalidomide and lenalidomide in relapsed/refractory MM patients. The emergence of these drugs has resulted in a clear improvement in the outcome of these patients in the last years, with an increase in median overall survival of up to five years.

Nevertheless, despite this clear progress, most patients (if not all) eventually relapse and the outcome of MM patients once they become refractory or ineligible to receive bortezomib or an IMID is quite poor with a survival inferior to one year.Therefore novel therapeutic options are still necessary for these relapsed or refractory patients. In this regard, several drugs that target specific mechanisms of the tumoral cells are currently being explored in the preclinical and clinical setting.(10) Some examples of the most promising of these targeted agents are second-generation proteasome inhibitors or immunomodulatory agents, deacetylase inhibitors (DACi), the kinesin spindle protein inhibitor filanesib and several monoclonal antibodies.

Pembrolizumab (MK-3475) Programmed cell death 1 (PD-1) axis function and mechanism of action of MK-3475 The programmed cell death 1 (PD-1) receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated T cells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions.

PD-1 and family members are type I transmembrane glycoproteins containing an Ig Variable-type (V-type) domain responsible for ligand binding and a cytoplasmic tail responsible for the binding of signaling molecules. The cytoplasmic tail of PD-1 contains two tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif (ITIM) and an immunoreceptor tyrosine-based switch motif (ITSM). Following T-cell stimulation, PD-1 recruits the tyrosine phosphatases, SHP-1 and SHP-2, to the ITSM motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3ζ, PKCθ, and ZAP70, which are involved in the CD3 T-cell signaling cascade.

PD-1 (encoded by the gene Pdcd1) is an immunoglobulin (Ig) superfamily member related to CD28 and CTLA-4 which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD-L2).The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from, that of CTLA-4, as both molecules regulate an overlapping set of signaling proteins. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T cells, B cells, T regs, and natural killer cells. Expression has also been shown during thymic development on CD4-CD8- (double negative) T cells, as well as subsets of macrophages and dendritic cells.(20) The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types including non-hematopoietic tissues and in various tumors. Both ligands are type 1 transmembrane receptors containing both IgV- and IgC-like domains in the extracelular region and contain short cytoplasmic regions with no known signaling motifs. Binding of either PD-L1 or PD-L2 to PD-1 inhibits T-cell activation triggered through the T-cell receptor. PD-L1 is expressed at low levels on various non-hematopoietic tissues, most notably on vascular endothelium; whereas PD-L2 is only detectably-expressed on antigen-presenting cells found in lymphoid tissue or chronic inflammatory environments. PD-L2 is thought to control immune T-cell activation in lymphoid organs, whereas PDL1 serves to dampen unwarranted T-cell function in peripheral tissues.Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. High expression of PD-L1 on tumor cells (and to a lesser extent of PD-L2) has been found to correlate with poor prognosis and survival in various cancer types, including RCC, pancreatic carcinoma, HCC, and ovarian carcinoma. Furthermore, PD-1 has been suggested to regulate tumor-specific T-cell expansion in patients with melanoma. The observed correlation of clinical prognosis with PD-L1 expression in multiple cancers suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

MK-3475 (previously known as SCH 900475) is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. This blockade enhances functional activity of the target lymphocytes to facilitate tumor regression and ultimately immune rejection.

* Clinical experience with MK-3475 Several clinical trials are being conducted in advanced melanoma, non-small cell lung cancer, head and neck cancer, urothelial tract cancer, triple negative breast cancer, gastric cancer, and hematologic malignancies (including smoldering multiple myeloma). A phase I trial in combination with lenalidomide and dexamethasone is now enrolling MM patients. .
* Rationale for using anti-PD1 MoAb as consolidation in MM PD-L1 is expressed on most MM plasma cells, and PD-L1 overexpression enhanced MM invasiveness and rendered tumor cells less susceptible to cytotoxic T-lymphocytes (CTLs). This effect was alleviated by anti-PD-L1 antibody treatment, demonstrating the importance of the PD-1/PD-L1 pathway in this process. In addition, a recent report demonstrated increased levels of PD-L1 on MM cells together with enhanced PD-1 expression on T cells with an "exhausted" phenotype. The immunosuppressive effects of myeloma are overcome by PD-L1 blockade.(32) A Phase 1 clinical trial conducted in advanced hematologic malignancies using CT-011, showed clinical responses in 6 of 17 patients including stable disease in MM patients.

Moreover, a recent experiment performed by our group showed that MM patients in serological complete remission but with residual disease have clear overexpression of the molecules in this pathway both in tumor cells and also T-lymphocytes. And that was very clear when compared with MM patients in immunophenotypic CR (that is without residual cells in the bone marrow by flow cytometry). This could be suggesting that this pathway may be responsible, at least partially, of the inability to eradicate the tumor cells in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Performance status (ECOG) ≤ 2.
* Patient is, in the Investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Patients previously diagnosed with MM according to the IMWG Criteria (Blood 2011) who are in good response (≥VGPR) but with persistent residual disease after the end of any therapy administered for a limited duration of time either at 1st or 2nd line of therapy.

Persistent disease is defined by either the presence of an M-Component by electrophoresis, positive immunofixation, abnormal FLC ratio or identification of pathological plasma cells by flow cytometry.

* At least 2 months for any non-transplant therapy or 3 months after ASCT, must relapse from the last dose of the previous treatment before being eligible to be included in the trial.
* Response must be confirmed to be stable between the end of the previous therapy and the initiation of the trial (see the time that must elapse in the previous criteria).

Stable is defined as: No change in response according to the IMWG Criteria between these determinations; No evidence of increase or decrease (> 25%) in M-component, provided the variation is > 0.5 mg/dl; No evidence of increase or decrease (> 25%) of the involved FLC, provided the ratio is abnormal and the absolute change is > 10 mg/dL; No evidence of increase or decrease (> 50%) of the percentage of pathological plasma cells by flow cytometry in the bone marrow provided the variation is > 0.5%; No positivization or negativization of the electrophoresis or IFE between these determinations.

In case of doubt, another determination separated at least 1 month after the last one is required to confirm the stability of the response, and this must be discussed with the DMC, prior to be eligible.

Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or other antibody or drug specifically targeting T cell co-stimulation).
* Known hypersensitivity to pembrolizumab or any of its excipients.
* Non-adequate hematological or biochemical parameters as specified below:

Hemoglobin < 8.0 g/dl. Platelets count < 75 x109/L without previous platelet transfusions in the last 7 days.

Neutrophils (ANC) <1 × 109/L without growth factor support (defined as no growth factor administration for at least 14 days prior to observation).

Aspartate transaminase (AST): > 2.5 x the upper limit range. Alanine transaminase (ALT): > 2.5 x the upper limit range. Total bilirubin: > 2 x the upper limit range. Creatinine clearance: < 30 mL/min (measured or calculated with the Cockcroft and Gault formula).

* Absence of recovery from any significant non-hematological toxicity derived from previous treatments. The presence of alopecia and NCI CTCAE grade < 2 symptomatic peripheral neuropathy is allowed.
* Pregnant or lactating women or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment. Female subjects of childbearing potential should have a negative urine or serum pregnancy prior to study registration and re-tested within 72 hours prior to receiving the first dose of study medication.
* Men and women of reproductive potential who are not using effective contraceptive methods (double barrier method, intrauterine device, oral contraception). Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Previous history of any other malignancy in the last 5 years (except basal cell carcinoma, skin epithelioma or carcinoma in situ of any site).
* More than 2 prior lines of therapy for MM.
* Previous allogeneic stem cell transplantation.
* Other relevant diseases or adverse clinical conditions:

Congestive heart failure or angina pectoris, myocardial infarction within 12 months before inclusion in the study.

Uncontrolled arterial hypertension or cardiac arrhythmias (i.e. requiring a change in medication within the last 3 months or a hospital admission within the past 6 months).

History of significant neurological or psychiatric disorders. Active infection. Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).

Uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism) (i.e. requiring relevant changes in medication within the last month, or hospital admission within the last 3 months).

Active autoimmune disease or a documented history of autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the trial.

* Patient is known to be HIV positive, Hepatitis B surface antigen-positive, has active hepatitis C infection or has active tuberculosis.
* Limitation of the patient's ability to comply with the treatment or follow-up protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of Pembrolizumab as measured by overall response rate manteinance | 2 years

SECONDARY OUTCOMES:
Safety will be evaluated by assessing toxicity related to pembrolizumab | 2 years
Efficacy as measured by minimal residual disease rate after two years of maintenance treatment with pembrolizumab | 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital 12 de octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital General Morales Messeguer, Murcia
  - Hospital General Universitario Morales Messeguer, Murcia
  - Clinica Universitaria de Navarra, Pamplona
  - Hoapital Clinico Universitario Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Clinico de Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Puig N, Corchete-Sanchez LA, Perez-Moran JJ, Davila J, Paino T, de la Rubia J, Oriol A, Martin-Sanchez J, de Arriba F, Blade J, Blanchard MJ, Gonzalez-Calle V, Garcia-Sanz R, Paiva B, Lahuerta JJ, San-Miguel JF, Mateos MV, Ocio EM. Pembrolizumab as Consolidation Strategy in Patients with Multiple Myeloma: Results of the GEM-Pembresid Clinical Trial. Cancers (Basel). 2020 Dec 3;12(12):3615. doi: 10.3390/cancers12123615. PMID 33287189